CLINICAL TRIAL: NCT03275831
Title: A Pilot Study to Investigate the Efficacy of PluroGel in Healing Venous and Mixed Aetiology Leg Ulcers
Brief Title: PluroGel on Wounds of Mixed Etiology
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R17-006; WWIC/2016/02 (Other: Welsh Wound Innovation Centre)
Record Dates: First submitted 2017-08-29; First posted 2017-09-08 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Venous Ulcer; Arterial Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrasite Gel (Active Comparator): Intrasite Gel is an effective method for hydrating dry necrotic and sloughy wounds. It is an amorphous gel that contains 85% water, and gently increases the moisture level within the wound, encouraging moist wound healing through autolytic debridement.
  Interventions: Device: Intrasite gel
- PluroGel Burn and Wound Dressing (Experimental): PluroGel contains a surfactant-based cleanser to assist wound debridement and cleansing
  Interventions: Device: PluroGel

INTERVENTIONS:
Device: PluroGel — Surfactant based gel
  Arms: PluroGel Burn and Wound Dressing
Device: Intrasite gel — Hydrogel
  Arms: Intrasite Gel

SUMMARY:
A randomized controlled study (RCT) to investigate the topical effectiveness of PluroGel in healing venous and mixed aetiology leg ulcers. Patients with venous and mixed aetiology leg ulcers will be identified from hospital outpatient clinics. Willing patients meeting the inclusion and exclusion criteria will be consented and assessed in line with standard care. Participants will be randomized at Week 2 to receive either topical PluroGel or Intrasite gel (an alternative topical hydrogel product) if inclusion criteria is met.

DETAILED DESCRIPTION:
This will be a pilot, randomized, controlled, multi-center trial to determine the effectiveness of PluroGel in the reduction of size of wounds and reduction of slough covering the wound surface compared with Intrasite Gel. The primary objectives will be to evaluate the effectiveness of PluroGel compared with Intrasite Gel in the reduction of size of venous leg ulcers or mixed venous arterial aetiology. Also the reduction in the percentage of slough covering the wound bed in both groups will be compared. The secondary objective will be to evaluate patient comfort, satisfaction and acceptance of the hydrogels along with staff feedback of both hydrogels. Patients with either a venous leg ulcer (VLU) or an mixed venous arterial aetiology (MAU) leg ulcer will be identified by the participant's health care provider and will be treated with PluroGel or Intrasite Gel. A total of 40 subjects will be enrolled to the study, 20 to each arm. These subjects will be recruited from patients receiving treatment for wounds at NHS outpatient clinic. Participants will be approached initially by the NHS care-giver and asked if interested in participating in research. If interested, participants will be asked to sign a permission to contact form for contact details to be given to a member of the research team who would then contact the participant to provide further information. A screening log will be kept of all patients who have been considered but who do not fulfill the criteria for entry. Patients will be randomized to either Plurogel and standard care or Intrasite Gel in conjunction with standard care, on an equal basis. Subjects will be eligible for randomization if during the first two weeks within the study the target wound has not reduced in surface area by 30% or more and there has been a less than 25% reduction in the cover of the wound bed with visible slough. Once the subject has completed 4-weeks of treatment, and the final visit, or the target ulcer has healed, whichever is soonest, then the subject has completed the study and the termination form will be completed. The Investigator will ensure that all CRF forms are completed and accurate. The study end date will be the date of the last subject's last visit. The CI and study sponsor, will comply with any safety reporting obligations for serious adverse device related events to the manufacturer, study sponsor, R&D Department(s) of the University Health Board(s) and the Ethics Committee, as defined in the applicable laws and regulations, and within the required timelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years old
* Patients with a non-healing venous leg ulcer or mixed aetiology ulcer.
* Duration of wound ≥ 6 weeks ≤ 5 years
* Wound is ≥ 1 cm2 ≤ 100cm2 no length longer than 10cm
* Presence of at least 25% visible slough within the wound bed
* The patient must be able to understand the study and provide written informed consent
* No clinical signs of infection

Exclusion Criteria:

* Known hypersensitivity to any of the wound dressings or compression bandaging to be used in the trial
* Current local or systemic antibiotics in the week prior to inclusion
* Clinically infected wound as determined by the presence of 3 or more of the following clinical signs: perilesional erythema, pain between two dressing changes, malodorous wound, abundant exudate and oedema.
* Prolonged treatment with immunosuppressive agents or high dose corticosteroids
* Patients who have a current illness or condition which may interfere with wound healing in the last 30 days (carcinoma, connective tissue disease, autoimmune disease or alcohol or drug abuse)
* Patients who have participated in a clinical trial on wound healing within the past month
* Patients with a known history of non-adherence with medical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Change in wound size | 4 weeks
  Comparison of change in wound surface area (cm2) over a 4 week assessment between baseline and final assessment in PluroGel treated group compared to Intrasite treated group.
Change in average percent reduction of slough in wound bed over 4 week treatment | 4 weeks
  Comparison of change in average percent reduction of slough present in the wound bed observed at baseline and over 4 week treatment period in PluroGel treated group compared to Intrasite treated group

SECONDARY OUTCOMES:
Patient evaluation | Up to 6 weeks
  Survey questions to report adherence to protocol of care, comfort, comparison with previous treatments, level of patient discomfort and pain during use of either PluroGel or Intrasite
Staff evaluation | Up to 6 weeks
  Survey to record staff feedback including ease of application and removal of both PluroGel and the comparator Intrasite.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Aneurin Bevan University Health Board, Newport, South Wales
  - Cardiff & Vale University Health Board, Cardiff, Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Callam MJ, Harper DR, Dale JJ, Ruckley CV. Arterial disease in chronic leg ulceration: an underestimated hazard? Lothian and Forth Valley leg ulcer study. Br Med J (Clin Res Ed). 1987 Apr 11;294(6577):929-31. doi: 10.1136/bmj.294.6577.929. PMID 3107659
- [Background] Connor-Ballard PA. Understanding and managing burn pain: Part 2. Am J Nurs. 2009 May;109(5):54-62; quiz 63. doi: 10.1097/01.NAJ.0000351510.77627.db. PMID 19411907
- [Background] Cullum N, Nelson EA, Fletcher AW, Sheldon TA. Compression for venous leg ulcers. Cochrane Database Syst Rev. 2000;(3):CD000265. doi: 10.1002/14651858.CD000265. PMID 10908469
- [Background] Gottrup F, Apelqvist J, Price P; European Wound Management Association Patient Outcome Group. Outcomes in controlled and comparative studies on non-healing wounds: recommendations to improve the quality of evidence in wound management. J Wound Care. 2010 Jun;19(6):237-68. doi: 10.12968/jowc.2010.19.6.48471. PMID 20551864
- [Background] Hunter RL, Luo AZ, Zhang R, Kozar RA, Moore FA. Poloxamer 188 inhibition of ischemia/reperfusion injury: evidence for a novel anti-adhesive mechanism. Ann Clin Lab Sci. 2010 Spring;40(2):115-25. PMID 20421622